CLINICAL TRIAL: NCT05910437
Title: Optimizing Treatments for Heart Failure During Hospitalization
Acronym: OPTICARD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr. Nicolas GIRERD, coordinating investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI115
Record Dates: First submitted 2023-04-28; First posted 2023-06-18 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Decompensated Heart Failure
Keywords: Decompensated heart failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hospitalized patient for decompensated heart failure — Describe the evolution of heart failure medications during hospitalization for decompensated heart failure.

SUMMARY:
Heart failure reaches 1.5 million people in France and is responsible for 200,000 hospitalizations per year.

Over the past ten years, new therapies have emerged (treatment of martial deficiency, Entresto, iSGLT2).

Hospitalization in a context of acute heart failure is a moment of choice in the history of the disease to introduce recommended treatments under closer supervision (clinical, biological) than in ambulatory, and allows a decrease in hospitalizations, morbidity and mortality.

The purpose of this study is to describe the introduction of heart failure drugs (including iSGLT2) in real-life settings in patients hospitalized for decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years
* Hospitalized (≥24h) for decompensated heart failure in cardiology.

Exclusion Criteria:

* Patient opposition participation in research and use of data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized (≥24h) patient for decompensated heart failure in cardiology between november 2021 and october 2022
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Prescription score | During hospitalisation for decompensated heart failure (up to 10 days)
  Prescription score, ranging from 0 to 10, each type of heart failure treatment (IEC/ARA2, Sacubitril, betablockers, SGLT2i, MRA) being evaluated on a scale of 2.

SECONDARY OUTCOMES:
serum concentration of creatinine | During hospitalisation for decompensated heart failure (up to10 days)
  Creatinine measured at admission and discharge
serum concentration of potassium | During hospitalisation for decompensated heart failure (up to 10 days)
  Potassium measured at admission and discharge
Concentration of hemoglobin | During hospitalisation for decompensated heart failure (up to 10 days)
  hemoglobin measured at admission and discharge
All cause Death | 6 months
Rate of hospitalization for heart failure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, MD-PhD, Study Chair — CHRU de NANCY
Locations (2):
- France (2):
  - Chr Metz Thionville, Ars-Laquenexy
  - CHRU de NANCY, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No